CLINICAL TRIAL: NCT00220246
Title: Clinical and Molecular Characterization of Familial Microsatellite Stable Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Other Study IDs: EOMSD2004
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Colorectal Neoplasms
Keywords: Hereditary colorectal cancer; Microsatellite instability; Chromosomal instability
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability; Chromosomal Instability

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Two major genetic pathways leading to colorectal carcinoma can well be distinguished; the 'suppressor pathway', which is characterized by inactivation of tumor-suppressor genes and the 'mutator pathway', which is characterized by microsatellite instability. The purpose of this study is to explore a third putative pathway; microsatellite and chromosome stable colorectal cancer where an alternative cancer-causative mechanism might play a role.

DETAILED DESCRIPTION:
Patients with familial colorectal cancer will be characterized with respect to family history, medical history and demographic characteristics. The histopathology of the tumors will be reviewed. Tumor specimens will be analysed on molecular defects.

ELIGIBILITY:
Inclusion Criteria:

- Colorectal cancer before the age of 51 years

Microsatellite stable tumor

Exclusion Criteria:

-

Max Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130
Dates: Start 2004-03; Study Completion 2008-09

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline Hoogerbrugge, MD, PhD, Principal Investigator — Department of Human Genetics, Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University, Nijmegen, Netherlands

REFERENCES:
- [Background] Chan TL, Curtis LC, Leung SY, Farrington SM, Ho JW, Chan AS, Lam PW, Tse CW, Dunlop MG, Wyllie AH, Yuen ST. Early-onset colorectal cancer with stable microsatellite DNA and near-diploid chromosomes. Oncogene. 2001 Aug 9;20(35):4871-6. doi: 10.1038/sj.onc.1204653. PMID 11521198
- [Background] Hawkins NJ, Tomlinson I, Meagher A, Ward RL. Microsatellite-stable diploid carcinoma: a biologically distinct and aggressive subset of sporadic colorectal cancer. Br J Cancer. 2001 Jan;84(2):232-6. doi: 10.1054/bjoc.2000.1554. PMID 11161382
- [Background] Georgiades IB, Curtis LJ, Morris RM, Bird CC, Wyllie AH. Heterogeneity studies identify a subset of sporadic colorectal cancers without evidence for chromosomal or microsatellite instability. Oncogene. 1999 Dec 23;18(56):7933-40. doi: 10.1038/sj.onc.1203368. PMID 10637503